CLINICAL TRIAL: NCT03231189
Title: Prospective Multicentric Study for the Diagnostic Performance of CArdiac MAgnetic REsonance Imaging Used First for the Diagnosis of Coronary Artery Disease as the Etiology of Left Ventricular Dysfunction
Brief Title: Cardiac MRI in Front Line for the Diagnosis of Coronary Artery Disease as the Etiology of Left Ventricular Dysfunction
Acronym: CAMAREC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 16181
Record Dates: First submitted 2017-06-27; First posted 2017-07-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Coronary artery disease; cardiac MRI; heart failure
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
When a patient is newly diagnosed of systolic dysfunction without obvious etiology (such as rhythmic, ischemic, or valvular disease), most of the time a coronary angiography is performed. In this situation, the investigators aim to evaluate a strategy with CMR as the front line exam, and invasive coronary angiography performed only in case of ischemic scar on CMR Additionally, a secondary analysis of the collected CMR images will be performed by the MIRACL.AI core lab (AP-HP, Paris) using artificial intelligence (AI) algorithms. This analysis aims to enhance the diagnostic accuracy of coronary artery disease (CAD) detection in patients with reduced left ventricular ejection fraction (rLVEF).

DETAILED DESCRIPTION:
Reduced Left Ventricular Ejection Fraction (LVEF) is estimated to be present in 3-7% of the population. With a survival rate between 25-40% at 5 years after a first hospitalization, prognosis of heart failure is similar to that of most cancers. Its treatment and prognosis strongly depend on the etiology, and coronary artery disease is the most frequent one. Identifying coronary artery disease determines care, including medical treatment (aspirin, statins) and revascularization strategies (stent implantation, coronary artery bypass grafting). Once an echocardiography has revealed an LV reduction, with no clear etiology at clinical or echographical examination, coronary angiography is almost systematically performed. But among the 260,000 invasive coronary angiographies performed each year in France (all indications included), 30-60% are "normal" (no obstructive coronary artery).

And among patients with unexplained LV dysfunction, this rate reaches 70-74%… Thus the efficiency of systematic coronary angiography is questionable for these latter. Besides, angiography is invasive, and associated with multiple risks and costs.

Cardiac Magnetic Resonance Imaging (CMR) is very specific and sensitive for detecting myocardial infarction. Small series concluded that a reduction of LVEF due to coronary artery stenosis should have at least one myocardial scar, detected on CMR. But the available data was not enough to change guidelines and clinical practice. In our retrospective study performed on 305 patients, the sensibility of CMR for coronary stenosis was 96%. Furthermore, CMR as a first-line exam would have avoided 71% of coronary angiography, saving 216 days of hospitalization and 329.054 € (1.079€/patient). These results reinforce the previous data but are not definitive.

The aim of this study is to provide a high level of evidence of the benefits and safety of a strategy based on CMR as the front line exam for newly diagnosed systolic dysfunctions.

The primary objective is to evaluate the sensitivity of CMR for predicting the presence of angiographically significant coronary artery stenosis in patients with reduced LVEF. The primary endpoint is the sensitivity of CMR for predicting the presence of significant coronary artery stenosis on coronary angiography in patients with reduced LVEF.

The objective of the economic evaluation is to estimate the incremental (or decremental) cost effectiveness of using CMR first compared to coronary angiography first.

As part of the secondary analysis, CMR images from the CAMAREC study will be transferred to the Multimodality Imaging for Research and Analysis Core Laboratory for Artificial Intelligence (MIRACL.AI) at AP-HP, Paris. The MIRACL.AI team, led by Dr. Theo Pezel, will apply advanced AI algorithms to detect ischemic patterns and quantify myocardial scarring. This AI analysis aims to improve the sensitivity and specificity of CMR in identifying significant CAD and non-ischemic cardiomyopathies.

For unexplained LV dysfunction, patient will be addressed for CMR first and coronary angiography within 2 weeks after (instead of systematic coronary angiography and unsystematic CMR). CMR and coronary angiography will be performed in all patients. Independent committees will blindly review CMRs and coronary angiographies at the end of the study.

Data from the CAMAREC study will be securely transferred to MIRACL.AI for AI-based analysis. This transfer does not affect the data flow to Lariboisière, nor the confidentiality or the study's timeline. MIRACL.AI will solely focus on the AI-enhanced interpretation of the CMR images.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Left Ventricular Ejection Fraction ≤ 45% on transthoracic echocardiography
* Informed signed consent
* Patient having had a preliminary clinical examination

Exclusion Criteria:

* Known significant coronary artery stenosis (history of myocardial infarction or coronary artery stenosis).
* Formal indication for coronary angiography other than LV dysfunction (typical angina, acute coronary syndrome, …).
* Obvious etiology for LV dysfunction (valvular, rhythmic…).
* Pregnancy or breastfeeding.
* Other contraindication for CMR (severe allergy to gadolinium known), or coronary artery angiography.
* First diagnosis of LVEF dysfunction > 8 weeks.
* Non covered patient by the social security, the CMU
* Patients under guardianship, or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred in one of the participating centers for the etiologic assessment of an unexplained LVEF reduction will be assessed for eligibility.
  A trans-thoracic echocardiography will be performed in the center at the inclusion as usual, to assess LVEF and confirm the absence of obvious explanation to its reduction.
  Standard biological tests (included in the standard biological investigation of dilated cardiomyopathy) will be performed to exclude any contraindications to coronary angiography as usual care. They are the same as those required before CMR.
Sampling Method: Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CMR for predicting the presence of significant coronary artery stenosis on coronary angiography in patients with reduced LVEF. | up to 8 weeks
  The primary endpoint is the sensitivity (and its 95% confidence interval) of CMR for the diagnosis of significant coronary artery stenosis on coronary angiography in patients with reduced LVEF.
  This sensitivity is the following ratio:
  Number of patients with an ischemic scar on CMR and a significant coronary artery stenosis on coronary angiography / Number of patients with a significant coronary artery stenosis on coronary angiography.

SECONDARY OUTCOMES:
Evaluation of the other diagnostic performances indices of CMR for the diagnosis of angiographically significant coronary artery stenosis in patients with reduced LVEF | up to 8 weeks
  Sensitivity¸ specificity, positive predictive value and negative predictive value (and their 95% confidence interval) of CMR for the diagnosis of significant coronary artery stenosis on coronary angiography in patients with reduced LVEF
Evaluation of the diagnostic performances of CMR for predicting angiographically significant coronary artery stenosis in patients with reduced LVEF requiring revascularization. | up to 8 weeks
  Sensitivity¸ specificity, positive predictive value and negative predictive value (and their 95% confidence interval) of CMR for the diagnosis of significant coronary artery stenosis on coronary angiography in patients with reduced LVEF requiring revascularization
Analysis of the concordance of CMR and coronary artery angiography in terms of coronary artery territory in patients with coronary stenosis. | up to 8 weeks
  κ concordance coefficient between CMR and coronary angiography for the diagnosis of affected myocardial territory in patients with coronary artery stenosis.
Additional value of CMR for the etiologic diagnosis of reduced LVEF including non-ischemic (LV non compaction, myocarditis …). | up to 8 weeks
  Proportion of different etiological diagnosis of reduced LVEF provided only by CMR
Additional value of CMR for the diagnosis of complications of reduced LVEF (LV thrombus mainly). | up to 8 weeks
  Number of patients for whom a complication due to LVEF reduction (LV thrombus, left ventricular dys-synchrony, pre-ruptured left ventricular wall...) is provided only by CMR.
Additional value of CMR for the decision of coronary artery revascularization. | up to 8 weeks
  Proportion of patients with coronary stenosis on the coronary angiography for whom CMR change the decision of revascularization, due to the absence of myocardial viability.
Evaluate the reproducibility of the interpretations of CMR for ischemic cardiomyopathy. | up to 8 weeks
  κ concordance coefficient between the first interpretation of CMR (in the participating centers), and the second (by the CMR reading committee).
AI-Based Diagnostic Performance of CMR | At the end of the study (43 months)
  The MIRACL.IA team will use advanced AI algorithms to detect ischemic patterns.
AI-Based Diagnostic Performance of CMR | At the end onf the study (43months)
  The MIRACL.AI team will apply advanced AI algorithms to quantify myocardial scarring

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Jondeau, MD,PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Bichat Claude-Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desroche LM, Darmon A, Lavie-Badie Y, Mandry D, Ducrocq G, Si-Moussi T, Durand-Zaleski I, Millischer D, Milleron O, Huttin O, Valla M, Mangin L, Farah B, Diakov C, Logeart D, Safar B, Travers JY, Mesnier J, Vappereau A, Alfaiate T, Burdet C, Jondeau G; CAMAREC investigators. Diagnostic accuracy of late gadolinium enhancement cardiac MRI for coronary artery disease in patients with reduced left ventricular ejection fraction. Heart. 2025 Sep 25;111(20):969-975. doi: 10.1136/heartjnl-2024-325419. PMID 40147871